CLINICAL TRIAL: NCT01619579
Title: Effects of a 4 Week AVACEN Treatment on Pain Perception in Fibromyalgia - An Open Label Study
Brief Title: Investigation of AVACEN Thermal Exchange System for Fibromyalgia Pain
Acronym: AVACEN: TES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avacen, Inc. (Industry)
Collaborators: University of California, San Diego (Other); San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110973
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Results first posted 2015-12-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pain; Non-Invasive; Arthritis; Rheumatoid Disease
MeSH Terms: conditions — Fibromyalgia; Pain; Arthritis | interventions — Microscopy, Electron, Transmission

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Subjects with Fibromyalgia undergo twice daily use of the non-invasive device for 4 weeks.
  Interventions: Device: AVACEN Thermal Exchange System

INTERVENTIONS:
Device: AVACEN Thermal Exchange System — Non-invasive device forms vacuum around subject's hand, enabling efficient core body temperature adjustment using heating element inside device.
  Other Names: AVACEN Treatment Method (ATM) (previously known as the AVACEN Thermal Exchange System [TES] or the AVACEN Thermal Exchange Method [TEM])

SUMMARY:
Hypothesis: Daily use of the AVACEN Thermal Exchange System for 4 weeks will show improved Fibromyalgia pain and functioning markers, as assessed by biomarkers and clinical and psychological assessment. This non-invasive device is able to rapidly raise the core body temperature of the user by placing a hand in a vacuum chamber and resting it upon a heating element. The change in body temperature may change the sympathetic nervous system's activity and thereby reduce Fibromyalgia pain.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia diagnosis
* Over the age of 18
* Understands English
* Not pregnant/planning to become pregnant
* Average pain of 4 or greater over the last week (10 point scale)
* Fibromyalgia pain lasting longer than 6 months

Exclusion Criteria:

* Pregnant/Planning to become pregnant
* Major unstable psychiatric illness
* Major, uncontrolled systemic illness for which you may be hospitalized in the next 6 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VA San Diego, La Jolla, California, United States

REFERENCES:
- See also: Device manufacturer's website — http://www.avacen.com
- See also: VA San Diego website. Location study is conducted. — http://www.sandiego.va.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The design and the associated protocols were approved by the Institutional Review Boards of the University of California San Diego and the U.S. Department of Veteran Affairs. Pre- and post-treatment evaluations were conducted at the UCSD Pain Medicine Clinic in San Diego, CA.
Pre-assignment Details: Participants enrolled were diagnosed with FMS according to the 2010 ACR diagnostic criteria and were advised to refrain from stopping, changing, or starting any new treatment programs other than the study intervention. Patients who recently started, stopped, or changed pain or mood treatment were ineligible to enroll until three months had elapsed.
Groups:
- Treatment Group A: Treatment Group A (n=5) underwent one AVACEN Treatment Method (ATM) warming session for 10 minutes daily.
- Treatment Group B: Treatment Group B (n=17) underwent two AVACEN Treatment Method (ATM) warming sessions for 15 minutes daily.
Period: Overall Study
Arm/Group | Treatment Group A | Treatment Group B
Started | 5 | 17
Completed | 5 | 14
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group A: Treatment Group A (n=5) underwent one AVACEN Treatment Method (ATM) warming session for 10 minutes daily. The participants completed the warming treatment sessions at home.
- Treatment Group B: Treatment Group B (n=17) underwent two AVACEN Treatment Method (ATM) warming sessions for 15 minutes daily. The participants completed the warming treatment sessions at home.
- Total: Total of all reporting groups
Arm/Group | Treatment Group A | Treatment Group B | Total
Number analyzed (Participants) | 5 | 17 | 22
Age, Customized [Mean (Full Range); unit: years]
  Age | 41 [21 to 62] | 52 [31 to 76] | 48 [21 to 76]
Gender [Count of Participants; unit: Participants]
  Female | 5 | 15 | 20
  Male | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 17 | 22
Widespread Pain Index (WPI) [Mean (Full Range); unit: units on a scale] — BASELINE SCORE DESCRIPTION:
  Widespread Pain Index (WPI) Score Range is 0 to 19 points. 0 = Lowest pain score (Best Outcome). 19 = Highest pain score (Worst Outcome). Full Baseline Range of Group A Results: 13 to 18 points. Full Baseline Range of Group B Results: 8 to 19 points. 15.4 was the Baseline Average WPI Score for Treatment Group A. 15.0 was the Baseline Average WPI Score for Treatment Group B. Widespread pain was defined as pain occurring in at least 2 contralateral body quadrants, in addition to the axial skeleton for at least 3 consecutive months.
  units on a scale | 15.4 [13 to 18] | 15.0 [8 to 19] | 15.1 [8 to 19]
Tender Point Count (TPC) [Mean (Full Range); unit: units on a scale] — BASELINE SCORE DESCRIPTION:
  Tender Point Count (TPC) Score Range is 0 to 18. 0 = Lowest pain score (Best Outcome). 18 = Highest pain score (Worst Outcome). The criteria required confirming tenderness used 4kg of pressure applied to a total of 18 specified tender point sites.
  Fibromyalgia is diagnosed with a minimum tenderness count in 11 of 18 points. Full Baseline Range of Group A Results: 12 to 18 points. Full Baseline Range of Group B Results: 6 to 18 points. 15.4 was the Baseline Average TPC Score for Group A. 14.07 was the Baseline Average TPC Score for Group B.
  units on a scale | 15.4 [12 to 18] | 14.07 [6 to 18] | 14.4 [6 to 18]
Symptom Severity (SS) Score [Mean (Full Range); unit: units on a scale] — BASELINE SCORE DESCRIPTION:
  Symptom Severity (SS) Score Range is 0 to 12. 0 = Lowest pain score (Best Outcome). 12 = Highest pain score (Worst Outcome).
  The SS scale identifies the level of severity sum of 4 categories (Fatigue, Waking Unrefreshed, Cognitive Symptoms, Somatic Symptoms) over the past week, using this scale:
  0 = no problem
  1. = slight or mild
  2. = moderate
  3. = severe: continuous, life-disturbing
  Full Baseline Range of Group A: 5 to 12 points. Full Baseline Range of Group B: 6 to 12 points. 9.0= Baseline Average for Group A. 9.3= Baseline Average for Group B.
  units on a scale | 9.0 [5 to 12] | 9.3 [6 to 12] | 9.2 [5 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Widespread Pain Index (WPI) Score After 4 Weeks Treatment
Description: Widespread Pain Index (WPI) Score Range is 0 to 19 points. 0 = Lowest pain score (Best Outcome). 19 = Highest pain score (Worst Outcome). Widespread pain was defined as pain occurring in at least 2 contralateral body quadrants, in addition to the axial skeleton for at least 3 consecutive months.
Time Frame: 4 Weeks
Population: Enrolled population was diagnosed with FMS according to the 2010 ACR diagnostic criteria. Three participants withdrew from the study for personal reasons and their post-therapy data were not obtained.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 5 | 14
units on a scale | 13.0 [8 to 17] | 8.9 [3 to 18]

2. Primary Outcome: Tender Point Count (TPC) After 4 Weeks Treatment
Description: Tender Point Count (TPC) Score Range is 0 to 18. 0 = Lowest pain score (Best Outcome). 18 = Highest pain score (Worst Outcome). The criteria required confirming tenderness used 4kg of pressure applied to a total of 18 specified tender point sites.
  Fibromyalgia is diagnosed with a minimum tenderness count in 11 of 18 points.
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 5 | 13
units on a scale | 12.6 [6 to 18] | 10.0 [2 to 18]

3. Primary Outcome: Symptom Severity (SS) Score After 4 Weeks Treatment
Description: Symptom Severity (SS) Score Range is 0 to 12. 0 = Lowest pain score (Best Outcome). 12 = Highest pain score (Worst Outcome).
  The SS scale identifies the level of severity sum of 4 categories (Fatigue, Waking Unrefreshed, Cognitive Symptoms, Somatic Symptoms) over the past week, using this scale:
  0 = no problem
  * slight or mild
  * moderate
  * severe: continuous, life-disturbing
Time Frame: 4 Weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Treatment Group A | Treatment Group B
Number analyzed (Participants) | 5 | 14
units on a scale | 8.4 [5 to 11] | 7.4 [4 to 11]

ADVERSE EVENTS:
Time Frame: 4-week data collection period: No adverse events related to use of the ATM device or the ATM warming therapy were reported by any of the participants during the study.
Description: No adverse events related to use of the ATM device or the ATM warming therapy were reported by any of the participants during the study.
Arm/Group | Treatment Group A | Treatment Group B
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/17
Other Adverse Events (participants affected / at risk) | 0/5 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days